CLINICAL TRIAL: NCT02631018
Title: Sisters in Health: A Weight Loss Study for African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Principal Investigator, Loneke T. Blackman Carr, Doctoral Candidate, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0484
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Enhanced Weight Loss Intervention (Experimental): Participants will engage in 18 weight loss intervention group sessions over 6 months. Sessions will occur weekly for the first 3 months, and biweekly for the latter 3 months. Participants will receive a behavioral weight loss curriculum, calorie and physical activity recommendations. This arm, uniquely, will receive a culturally based physical activity component.
  Interventions: Behavioral: Physical Activity Enhanced Weight Loss Intervention
- Standard Weight Loss Intervention (Active Comparator): Participants will engage in 18 weight loss intervention group sessions over 6 months. Sessions will occur weekly for the first 3 months, and biweekly for the latter 3 months. Participants will receive a behavioral weight loss curriculum, calorie and physical activity recommendations.
  Interventions: Behavioral: Standard Weight Loss Intervention

INTERVENTIONS:
Behavioral: Standard Weight Loss Intervention — 18 session, group-based, 6-month, standard behavioral weight loss intervention
  Arms: Standard Weight Loss Intervention
Behavioral: Physical Activity Enhanced Weight Loss Intervention — 18 session, group-based, 6-month, physical activity enhanced behavioral weight loss intervention
  Arms: Physical Activity Enhanced Weight Loss Intervention

SUMMARY:
The purpose of this study is to compare the effect of a physical activity-enhanced behavioral weight loss intervention, compared to a standard behavioral weight loss intervention in African American women.

DETAILED DESCRIPTION:
A disparity exists in the prevalence of overweight and obesity between non-Hispanic white (NHW) and African American (AA) women. More AA women (78.2%) are overweight or obese compared to NHW (61.2%). Obesity increases the risk of developing numerous chronic diseases, including type 2 diabetes (T2DM), hypertension, cardiovascular disease, and some cancers. Among AA women, there is a higher prevalence, and almost double the risk, of developing T2DM compared to NHW. African Americans also have higher rates of complications and mortality from T2DM, and are more at risk for hypertension compared to NHW. Obesity is a costly epidemic. Fortunately, weight is a modifiable risk factor for reducing or preventing obesity and related diseases.

Interventions to reduce overweight and obesity through lifestyle change have been less effective for AA women compared to NHW women. African American women tend to lose less weight in standard behavioral weight loss interventions. A potential reason for smaller weight loss is that compared to NHW women, AA women have been shown to engage in less physical activity (PA) during these interventions.

The Sisters in Health study will test the efficacy of a 6-month randomized controlled trial in overweight and obese African American women. Women will be recruited to participate in this study comparing a standard behavioral weight loss intervention (BWI) to a physical activity enhanced BWI (BWI-PA) for 6 months. The primary objective of this study is to determine if AA women randomized to the BWI-PA will experience greater weight loss and PA compared to women receiving the BWI. Women in both groups will receive 18 face-to-face sessions on a tapered basis (weekly to biweekly). Face-to-face sessions will provide women with the knowledge, behavioral skills and strategies for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years old
* Ability to read, write, and speak English

  * Female gender
  * African American/Black/African/Afro-Caribbean race (self-identified)
  * BMI 25-45 (> 45 may have greater risks while participating)
  * Meets criteria for low active (defined as <3 days/week of at most 20 min. of PA/day) assessed by X
  * Willingness to be randomized
  * Willingness to participate for 6 months, including attending face-to-face sessions & outside of session tasks
  * Access to a computer reliable internet access
  * Willingness to use an app for diet and physical activity monitoring
  * Regularly used email address
  * Not planning to relocate
  * Able to attend group sessions on scheduled day

Exclusion Criteria:

* Recently lost weight, 5-10% in last 6 months
* Currently participating in another weight loss or PA study, or taking weight loss medication, and unwilling to discontinue those activities
* Pregnant or planning to become pregnant
* Any physical limitations to engaging in or increasing physical activity/exercise- assessed by PAR-Q (including but not limited to heart attack/myocardial infarction, congestive heart failure)
* Type 2 diabetes being treated with insulin
* Major psychological disorder
* History of diagnosed eating disorder
* Medications that affect weight (determined by study staff)

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F. Tate, PhD, Study Chair — University of North Carolina, Chapel Hill; Loneke T. Blackman Carr, MA, RD, Principal Investigator — University of North Carolina, Chapel Hill